CLINICAL TRIAL: NCT03955965
Title: OPTICONCIL: Implementation of Medication Reconciliation Process in an Emergency Department : Which Patients Should be Prioritized and How to Optimize Patients' Therapeutics?
Brief Title: Medication Reconciliation in an Emergency Department: How to Prioritize Patients ?
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: OPTICONCIL
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Emergency Service, Hospital; Medication Reconciliation
MeSH Terms: conditions — Emergencies | interventions — Medication Reconciliation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency patients with medication reconciliation: All patients who beneficiated from medication reconciliation in the emergency department between November 2017 and April 2018
  Interventions: Other: Medication reconciliation

INTERVENTIONS:
Other: Medication reconciliation — No intervention was performed other than collecting data on patients' medical files

SUMMARY:
Medication reconciliation has proven its efficiency in improving patients' care, especially for emergency patients.

This study aimed to identify risk factors of unintended medication discrepancies (UMD) in an emergency department. Secondary objectives were to identify the number and type of UMD, correction rate of UMD and the impact of emergency department organisation on UMD.

DETAILED DESCRIPTION:
Emergency patients are at high risk of medication errors, for different reasons: emergency admission, patients who don't know their at-home treatment (polymedicated, cognitive disorders, etc) and who don't have their medical prescriptions available.

Medication reconciliation has proven its efficiency in improving patients' care, especially for emergency patients. However, prioritization is essential to ensure a better efficiency of pharmaceutical resources.

In our center, a pharmacy resident has been assigned to medication reconciliation in the emergency department since November 2017, in collaboration with a clinical pharmacist. Every morning, 3 to 4 patients benefit from medication reconciliation (patients who will be transfered to another unit within our hospital).

The main objective was to identify risk factors of unintended medication discrepancies (UMD) in order to prioritize patients who will benefit from this newly implemented activity.

Secondary objectives were to identify the number and type of UMD, correction rate of UMD and the impact of emergency department organisation on UMD.

All patients who beneficiated from medication reconciliation in the emergency department between November 2017 and April 2018 were included. Were not included patients with a medication reconciliation performed but transfered to another hospital right after the emergency department visit.

This was a retrospective, monocentric, observational study. Number of patients required was 200. Variables collected were:

* demographics (age, sex, lifestyle, comorbidities),
* emergency care variables (date and time of medical care beginning, ambulance arrival, adressing type, medical prescriptions availability, main diagnosis, date and hour of medical prescriptions in the emergency department, prescriber (pharmacy/doctor), destination unit of patients)
* organizational variables (number of daily emergency visits, number of patients hospitalized within the emergency department),
* medical notes information on at-home treatment (number of missing information, of incorrect information, number of prescriptions in at-home treatment)
* medication reconciliation variables (date of medication reconciliation, number of sources of information needed, number of actual prescriptions in at-home treatment, number of intended medication discrepancies, number and type of UMD, time needed for medication reconciliation).

ELIGIBILITY:
Inclusion Criteria:

* All patients who beneficiated from medication reconciliation in the emergency department between November 2017 and April 2018

Exclusion Criteria:

* Patients transfered to another hospital right after the emergency department visit

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who beneficiated from medication reconciliation in the emergency department between November 2017 and April 2018
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Variables influencing the number of UMD in the emergency department | Nov2017-Apr2018
  Variation of the number of UMD for each variable was measured to identify the impact of each factor on medication errors (linear regression). Variables measured were the variables described in the protocol section.

SECONDARY OUTCOMES:
Number and type of UMD | Nov2017-Apr2018
Correction rate of UMD | Nov2017-Apr2018
Impact of organizational variables on the number of UMD | Nov2017-Apr2018

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Corny, PharmD, Principal Investigator — Pharmacy Department
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No